CLINICAL TRIAL: NCT01114568
Title: A Phase 1, Cross-Over, Single-Dose, Open-Label Study To Estimate The Relative Bioavailability Of Three Different Formulations Of PF-04971729 in Lean To Obese, Otherwise Healthy Adult Subjects
Brief Title: Study To Estimate The Relative Bioavailability of Ertugliflozin (PF-04971729, MK-8835) in Healthy Adult Participants (MK-8835-039)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 8835-039
Record Dates: First submitted 2010-04-27; First posted 2010-05-03 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Relative Bioavailability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — ertugliflozin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Ertugliflozin 10 mg: tablet→osmotic capsule (OC) fast→OC slow (Experimental): The three treatments are A) a single dose of 10 mg administered as 2x5 mg material sparing formulation tablets B) a single dose of 10 mg extemporaneously prepared osmotic capsule with target release rate of approximately 6 hours (EP-Osmotic Capsule-Fast) and C) a single dose of 10 mg extemporaneously prepared osmotic capsule with target release rate of approximately 14 hours (EP-Osmotic Capsule-Slow). Treatment are administered on Day 1, Hour 0 of each dosing period with a minimum of 7-days wash-out between treatments A, B, and C.
  Interventions: Drug: Ertugliflozin 10 mg tablet; Drug: Ertugliflozin OC Fast; Drug: Ertugliflozin OC Slow
- Ertugliflozin 10 mg: tablet→OC slow→OC fast (Experimental): The three treatments are A) a single dose of 10 mg administered as 2x5 mg material sparing formulation tablets B) a single dose of 10 mg EP-Osmotic Capsule-Fast and C) a single dose of 10 mg EP-Osmotic Capsule-Slow. Treatment are administered on Day 1, Hour 0 of each dosing period with a minimum of 7-days wash-out between treatments A, B, and C.
  Interventions: Drug: Ertugliflozin 10 mg tablet; Drug: Ertugliflozin OC Fast; Drug: Ertugliflozin OC Slow
- Ertugliflozin 10 mg: OC fast→tablet→OC slow (Experimental): The three treatments are A) a single dose of 10 mg administered as 2x5 mg material sparing formulation tablets B) a single dose of 10 mg EP-Osmotic Capsule-Fast and C) a single dose of 10 mg EP-Osmotic Capsule-Slow. Treatment are administered on Day 1, Hour 0 of each dosing period with a minimum of 7-days wash-out between treatments A, B, and C.
  Interventions: Drug: Ertugliflozin 10 mg tablet; Drug: Ertugliflozin OC Fast; Drug: Ertugliflozin OC Slow
- Ertugliflozin 10 mg: OC fast→OC slow→tablet (Experimental): The three treatments are A) a single dose of 10 mg administered as 2x5 mg material sparing formulation tablets B) a single dose of 10 mg EP-Osmotic Capsule-Fast and C) a single dose of 10 mg EP-Osmotic Capsule-Slow. Treatment are administered on Day 1, Hour 0 of each dosing period with a minimum of 7-days wash-out between treatments A, B, and C.
  Interventions: Drug: Ertugliflozin 10 mg tablet; Drug: Ertugliflozin OC Fast; Drug: Ertugliflozin OC Slow
- Ertugliflozin 10 mg: OC slow→tablet→OC fast (Experimental): The three treatments are A) a single dose of 10 mg administered as 2x5 mg material sparing formulation tablets B) a single dose of 10 mg EP-Osmotic Capsule-Fast and C) a single dose of 10 mg EP-Osmotic Capsule-Slow. Treatment are administered on Day 1, Hour 0 of each dosing period with a minimum of 7-days wash-out between treatments A, B, and C.
  Interventions: Drug: Ertugliflozin 10 mg tablet; Drug: Ertugliflozin OC Fast; Drug: Ertugliflozin OC Slow
- Ertugliflozin 10 mg: OC slow→OC fast→tablet (Experimental): The three treatments are A) a single dose of 10 mg administered as 2x5 mg material sparing formulation tablets B) a single dose of 10 mg EP-Osmotic Capsule-Fast and C) a single dose of 10 mg EP-Osmotic Capsule-Slow. Treatment are administered on Day 1, Hour 0 of each dosing period with a minimum of 7-days wash-out between treatments A, B, and C.
  Interventions: Drug: Ertugliflozin 10 mg tablet; Drug: Ertugliflozin OC Fast; Drug: Ertugliflozin OC Slow

INTERVENTIONS:
Drug: Ertugliflozin 10 mg tablet — A single dose of 10 mg ertugliflozin administered as 2x5 mg material sparing formulation tablets.
Drug: Ertugliflozin OC Fast — Formulation B) Ertugliflozin 10 mg OC Fast
Drug: Ertugliflozin OC Slow — Formulation C) Ertugliflozin 10 mg OC Slow

SUMMARY:
The purpose of this study is to examine the rate and extent of absorption of three oral formulations of ertugliflozin (PF 04971729, MK-8835) administered in lean to obese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 65 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests). Women must be of non childbearing potential
* Body Mass Index (BMI) of 18.5 to 35.4 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of screening).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen at Screening or prior to dosing in Period 1.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time 0 to time of the last quantifiable concentration (AUClast) for ertugliflozin | Up to 48 hr. postdose (Up to Day 3 in each dosing period)
AUC from Hour 0 to infinity (AUCinf) for ertugliflozin | Up to 48 hr. postdose (Up to Day 3 in each dosing period)
Maximum plasma concentration (Cmax) of ertugliflozin | Up to 48 hr. postdose (Up to Day 3 in each dosing period)
Time taken to reach the maximum observed plasma concentration (Tmax) of ertugliflozin | Up to 48 hr. postdose (Up to Day 3 in each dosing period)
Ertugliflozin half life (t1/2) | Up to 48 hr. postdose (Up to Day 3 in each dosing period)
Number of Participants Experiencing an Adverse Event (AE) | Up to 28 days postdose (Up to 49 days)
Number of Participants Discontinuing Study Drug Due to an AE | Up to Day 21
Urinary glucose excretion | Up to 48 hr. postdose (Up to Day 3 in each dosing period)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Marshall JC, Liang Y, Sahasrabudhe V, Tensfeldt T, Fediuk DJ, Zhou S, Krishna R, Dawra VK, Wood LS, Sweeney K. Meta-Analysis of Noncompartmental Pharmacokinetic Parameters of Ertugliflozin to Evaluate Dose Proportionality and UGT1A9 Polymorphism Effect on Exposure. J Clin Pharmacol. 2021 Sep;61(9):1220-1231. doi: 10.1002/jcph.1866. Epub 2021 Jun 19. PMID 33813736